CLINICAL TRIAL: NCT05892588
Title: Prevalence Study of Cardiovascular Diseases in a Population ≥ 65 Years in Italy
Acronym: PREVASC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Sponsor
Other Study IDs: PREVASC
Record Dates: First submitted 2023-05-25; First posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Valvular Heart Disease; Mitral Valve Disease; Aortic Valve Stenosis; Aortic Valve Insufficiency; Tricuspid Regurgitation
MeSH Terms: conditions — Heart Valve Diseases; Aortic Valve Stenosis; Aortic Valve Insufficiency; Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This registry is a large-scale epidemiological study (PREVASC) aimed at estimating the prevalence of symptomatic and asymptomatic valvular hear disease in men and women aged over 65 years randomly selected in Italy.

DETAILED DESCRIPTION:
PREVASC is a cross-sectional, population-based study. Participating subjects are invited from the general population and underwent a physical examination and an electrocardiography and echocardiographic examination by a local cardiologist. A random sample of about 2000 subjects over 65 years will be considered for sampling. The sample size is determined on the basis of a priori criteria in order to estimate a prevalence of 3% [standard error (SE) ± 1.1] for VHD.

Both clinical and demographic information will be collected to better characterize the invited population. Written informed consent for the clinical examination will be asked.

Demographic variables, cardiovascular (CV) risk, clinical history, physical findings, and medications will be recorded in a Case Report Form (CRF) by physicians or trained nurses. Assessment of anthropometric measures, blood pressure, and heart rate will be performed according to MONICA recommendations. Overweight is defined as a body mass index (BMI) between 25 and 29.9 kg/m2. Obesity is defined as BMI ≥30 kg/m2. Symptoms and signs attributable to VHD will be evaluated and reported on the CRF by a dedicated expert physician in each site at the time of the physical examination.

Echocardiography Complete Colour Doppler echocardiography will be performed in peripheral centers using commercially available machines according to a pre-defined protocol. Echocardiograms will be recorded in standard DICOM format on digital.

The following parameters will be acquired:

* Linear measurements of cardiac chambers will be obtained from the two-dimensional (2D) parasternal long axis view or, when available, from the M-mode parasternal short axis recording according to the recommendations of the European American Society of Echocardiography and the European Association of Cardiovascular Imaging [].
* LV volumes will be obtained from the apical four-chamber view and the EF calculated by using the modified Simpson's rule method.
* Left ventricular mass will be calculated according to the Devereux formula.
* Left ventricular systolic function will be calculated using the formula for ejection fraction EF: EDV-ESV/EDV X100.
* Also left atrium area or volume will be measured by the 4-chamber view.
* Calcifications of the aortic valve and mitral apparatus will be quantified as light, moderate, or severe, according to a published approach. The bicuspid aortic valve will be searched for and recorded. Trans-aortic and trans-mitral gradients, as well as mitral, aortic, and tricuspid regurgitation, will be reported and quantified according to continuous wave Doppler and Color Doppler area of regurgitation or vena contracta (VC) width (light, moderate, severe), respectively. For quantitative measurement of mitral regurgitation and tricuspidal regurgitation PISA method will be used. For aortic regurgitation PHT will be adopted other than VC. The aortic valve area will be calculated using the continuity equation other than the planimetric area. Mitral valve area will be calculated using pressure half time (PHT) other than planimetric area. Pulmonary artery systolic pressure will be estimated according to standard method.
* Doppler-derived indexes of transmitral flow and pulmonary vein flow, and tissue Doppler imaging of the lateral mitral annulus (E/e') will be used to define diastolic LVD. Peak early diastolic filling wave (E) velocity, peak atrial diastolic filling wave (A) velocity, and deceleration time of the E wave (DTE) will be measured at the tips of the mitral leaflets. The DTE will be calculated as the time from E to the time when the descent of E intercepts the zero line. The duration of the transmitral A wave velocity will also be measured. The peak velocity of pulmonary venous (PV) systolic (S), and diastolic (D) flow, the peak velocity of PV backward flow at atrial contraction (PVa), and the PVa wave duration (PVa dur) will be measured with the sample volume placed in the right upper pulmonary vein in the four-chamber axis view. The difference between the transmitral A wave duration (Adur) and PVa dur will be derived as an indirect index of increased LV filling pressures, according to the standard method. Tissue Doppler will be used to calculate the E/e' ratio.
* All digital echocardiograms will be analyzed offline on a dedicated workstation by three independent observers, blind to clinical data, and reviewed by the same experienced reader. Measurements will be expressed as an average of three cycles in sinus rhythm and from three to five cycles in atrial fibrillation.

Cardiologists and nurses will be trained locally according to standardized methodologies. Before enrolment begins, all participating centers will be required to perform and send an echo test to the Core Lab to verify the appropriateness of the acquisition procedure.

ELIGIBILITY:
Inclusion Criteria:

* All subject ≥ 65 years with no history of previous valvular heart disease

Exclusion Criteria:

* Age <65 years
* Any acute disease
* Recent hospitalization (until 1 month).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Subject with > 65 years with no history of previous valvular heart disease living in villages with less than 3000 inhabitants.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-05-07 (Actual); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
VALVOLAR HEART DISEASE PREVALENCE | at baseline
  The aim is to estimate the prevalence of symptomatic and asymptomatic valvolar heart disease in men and women aged over 65 years randomly selected in Italy: a complete colour-Doppler echocardiography will be performed in peripheral centres using commercially available machines according to a pre-defined protocol. Echocardiograms will be recorded with standard DICOM format on digital

SECONDARY OUTCOMES:
LEFT VENTRICOLAR DIMENSIONS AND FUNCTION | at baseline
  The aim is to estimate the prevalence of symptomatic and asymptomatic valvular heart disease in men and women aged over 65 years randomly selected in Italy: complete colour-Doppler echocardiography will be performed in peripheral centers using commercially available machines according to a pre-defined protocol. Echocardiograms will be recorded in standard DICOM format on digital
BURDEN OF ATRIAL FIBRILLATION | baseline
  The aim is to assess the burden of atrial fibrillation: a 12-lead electrocardiogram is performed to all patients enrolled

CONTACTS AND LOCATIONS:
Locations (1):
- AOUCareggi, Florence, Italy